CLINICAL TRIAL: NCT01225315
Title: A Multi-center, Double-blind, Placebo-controlled, Parallel-group Study to Establish Proof-of-concept and Explore the Efficacy of Different Doses of ACT-129968 in Adult Patients With Partly Controlled Asthma
Brief Title: Clinical Study to Explore the Efficacy of ACT-129968 in Patients With Partly Controlled Asthma
Acronym: CONTROL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-060A202
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — 2-(2-(1-naphthoyl)-8-fluoro-3,4-dihydro-1H-pyrido(4,3-b)indol-5(2H)-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Setipiprant - Dose 1 (Experimental): 100 mg b.i.d.
  Interventions: Drug: Setipiprant
- Setipiprant - Dose 2 (Experimental): 500 mg b.i.d.
  Interventions: Drug: Setipiprant
- Setipiprant - Dose 3 (Experimental): 1,000 mg b.i.d
  Interventions: Drug: Setipiprant
- Matching Placebo (Placebo Comparator): Oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching placebo administered orally twice daily
  Other Names: matching placebo
  Arms: Matching Placebo
Drug: Setipiprant — ACT-129968 (Dose 1, Dose 2, or Dose 3) administered orally twice daily
  Other Names: ACT-129968
  Arms: Setipiprant - Dose 1; Setipiprant - Dose 2; Setipiprant - Dose 3

SUMMARY:
This study will assess the efficacy and safety of ACT-129968 in subjects with partly controlled asthma on reliever therapy only.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* Males and females age 18 to 65 years
* Women of childbearing potential must use adequate contraception
* Presenting with a diagnosis of asthma according to GINA Guidelines
* Pre-bronchodilator forced expiratory volume in one second (FEV1) < / = 85% of patient's predicted normal value
* Reversibility of airway obstruction of > / = 12% and > / = 200mL from pre-bronchodilator FEV1
* ACQ score > / = 1.5

Exclusion Criteria:

* History of life-threatening asthma
* Any asthma exacerbation requiring treatment with systemic corticosteroids within the last 3 months
* Ongoing or recent treatment with medication for allergic airway disease
* Smoking within the last year, or life-time consumption > / = 10 pack-years (e.g., 20 cigarettes/day for 10 years)
* History of chronic pulmonary disease (other than asthma), such as chronic obstructive pulmonary disease (COPD), fibrosis, tuberculosis or sarcoidosis
* Pregnant or lactating women
* Diagnosis of aspirin or non-steroidal anti-inflammatory drug (NSAID)-induced asthma
* Any hospital admission for asthma within the last 6 months
* Anti-IgE therapy at any time check/update interventions by explicitely writing the experimental drug dosage in the interventions description
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2010-11-01; Primary Completion 2012-01-01 (Actual); Study Completion 2012-02-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate a change in forced expiratory volume while taking ACT-129968 versus placebo | Baseline to week 12

SECONDARY OUTCOMES:
Explore the efficacy of different doses of ACT-129968 on change in lung function and asthma control | Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mangialaio, MD, Study Director — Actelion
Locations (97):
- United States (22):
  - Clinical Investigative Site # 6204, Los Angeles, California
  - Clinical Investigative Site 6208, Los Angeles, California
  - Clinical Investigative Site # 6219, Tallahassee, Florida
  - Clinical Investigative Site 6213, Normal, Illinois
  - Clinical Investigative Site # 6215, New Orleans, Louisiana
  - Clinical Investigative Site # 6211, North Dartmouth, Massachusetts
  - Clinical Investigative Site # 6209, St Louis, Missouri
  - Clinical Investigative Site 6205, The Bronx, New York
  - Clinical Investigative Site # 6223, Winston-Salem, North Carolina
  - Clinical Inverstigative Site #6201, Lake Oswego, Oregon
  - Clinical Investigative Site # 6207, Medford, Oregon
  - Clinical Investigative Site # 6214, Portland, Oregon
  - Clinical Investigative Site 6203, Philadelphia, Pennsylvania
  - Clinical Investigative Site # 6228, Greenville, South Carolina
  - Clinical Investigative Site 6230, Spartanburg, South Carolina
  - Clinical Investigative Site 6202, Knoxville, Tennessee
  - Clinical Investigative Site 6226, Nashville, Tennessee
  - Clinical Investigative Site # 6220, El Paso, Texas
  - Clinical Investigative Site # 6225, Fort Worth, Texas
  - Clinical Investigative Site # 6222, San Antonio, Texas
  - Clinical Investigative Site 6229, San Antonio, Texas
  - Clinical Investigative Site # 6217, Madison, Wisconsin
- Australia (3):
  - Clinical Investigative Site 5002, Glebe
  - Clinical Investigative Site 5003, Nedlands
  - Clinical Investigative Site 5001, Sherwood
- Bulgaria (4):
  - Clinical Investigative Site # 5103, Rousse
  - Clinical Investigative Site # 5101, Sofia
  - Clinical Investigative Site # 5104, Sofia
  - Clinical Investigative Site # 5102, Stara Zagora
- Germany (8):
  - Clinical Investigative Site 5208, Berlin
  - Clinical Investigative Site 5212, Berlin
  - Clinical Investigative Site 5205, Dortmund
  - Clinical Investigative Site 5207, Gelnhausen
  - Clinical Investigative Site 5211, Hamburg
  - Clinical Investigative 5209, Lübeck
  - Clinical Investigative Site 5204, Mainz
  - Clinical Investigative Site 5202, Rüdersdorf
- Hungary (9):
  - Clinical Investigative Site 5310, Budapest
  - Clinical Investigative Site 5307, Csorna
  - Clinical Investigative Site 5304, Miskolc
  - Clinical Investigative Site # 5303, Nyíregyháza
  - Clinical Investigative Site 5309, Sátoraljaújhely
  - Clinical Investigative Site 5301, Siófok
  - Clinical Investigative Site # 5308, Sopron
  - Clinical Investigative Site # 5305, Szombathely
  - Clinical Investigative Site 5302, Tatabánya
- Israel (7):
  - Clinical Investigative Site # 5407, Ashkelon
  - Clinical Investigative Site 5401, Haifa
  - Clinical Investigative Site # 5402, Jerusalem
  - Clinical Investigative Site 5405, Petach Tikvah
  - Clinical Investigative Site # 5403, Rehovot
  - Clinical Investigative Site # 5404, Tel Aviv
  - Clinical Investigative Site # 5406, Tel Aviv
- Poland (5):
  - Clinical Investigative Site # 5507, Bialystok
  - Clinical Investigative Site # 5505, Krakow
  - Clinical Investigative Site # 5501, Lodz
  - Clinical Investigative Site # 5502, Lublin
  - Clinical Investigative Site # 5503, Tarnów
- Russia (10):
  - Clinical Investigative Site 5610, Barnaul
  - Clinical Investigative Site 5606, Barnaul
  - Clinical Investigative Site 5603, Kazan'
  - Clinical Investigative Site 5602, Moscow
  - Clinical Investigative Site 5654, Moscow
  - Clinical Investigative Site 5607, Moscow
  - Clinical Investigative Site 5609, Novosibirsk
  - Clinical Investigative Site 5605, Saint Petersburg
  - Clinical Investigative Site 5604, Saint Petersburg
  - Clinical Investigative Site 5608, Tomsk
- Serbia (2):
  - Clinical Investigative Site 5701, Belgrade
  - Clinical Investigative Site 5702, Belgrade
- Clinical Investigative Site 5802, Singapore, Singapore
- South Africa (9):
  - Clinical Investigative Site 5908, Bloemfontein
  - Clinical Investigative Site 5905, Cape Town
  - Clinical Ivestigative Site 5902, Cape Town
  - Clinical Investigative Site 5901, Durban
  - Clinical Investigative Site 5909, George
  - Clinical Investigative Site 5906, Johannesburg
  - Clinical Investigative Site 5910, Port Elizabeth
  - Clinical Investigative Site 5903, Pretoria
  - Clinical Investigative Site 5907, Pretoria
- Sweden (7):
  - Clinical Investigative Site 6001, Gothenburg
  - Clinical Investigative Site # 6006, Härnösand
  - Clinical Investigative Site 6003, Linköping
  - Clinical Investigative Site # 6002, Luleå
  - Clinical Investigative Site 6052, Lund
  - Clinical Investigative Site 6007, Stockholm
  - Clinical Investigative Site 6004, Varberg
- Ukraine (10):
  - Clinical Investigative Site # 6104, Donetsk
  - Clinical Investigative Site 6110, Kharkiv
  - Clinical Investigative Site # 6101, Kharkiv
  - Clinical Investigative Site # 6102, Kyiv
  - Clinical Investigative Site # 6103, Kyiv
  - Clinical Ivestigative Site 6111, Odesa
  - Clinical Investigative Site 6108, Poltava
  - Clinical Investigative Site # 6107, Uzhhorod
  - Clinical Investigative Site 6105, Zaporizhia
  - Clinical Investigative Site # 6106, Zaporizhia